CLINICAL TRIAL: NCT04434781
Title: Gastric Per-Oral Endoscopic Myotomy (G-POEM) for the Treatment of Gastroparesis: A Database Repository
Brief Title: Gastric Per-Oral Endoscopic Myotomy (G-POEM) for the Treatment of Gastroparesis
Acronym: G-POEM
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mohammad Al-Haddad, Associate Professor of Medicine, Associate Clinical Director, Indiana University
Other Study IDs: 1708840627
Record Dates: First submitted 2018-10-10; First posted 2020-06-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Gastroparesis
Keywords: GPOEM; Gastric Per-Oral Endoscopic Myotomy; Myotomy; Gastroparesis; g-poem
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastric Per-Oral Endoscopic Myotomy (G-POEM) is a procedure for the Treatment of Gastroparesis.

DETAILED DESCRIPTION:
Gastroparesis is a disease of the stomach where there is significant delay in gastric emptying of contents to the intestines. This disease results in a multitude of symptoms including nausea, vomiting, weight loss, and malnutrition.

Current treatments for gastroparesis include dietary changes, oral medications (prokinetic agents to enhance gastric motility, acid reducers, anti-emetics to reduce nausea and vomiting), gastric stimulators and rarely surgery.

G-POEM (Gastric Per-Oral Endoscopic Myotomy-creating a cut in the muscle that controls gastric emptying), an incision-less (no cutting of the surface of the body) endoscopic procedure, is increasingly being performed to assist in the management of certain groups of patients with gastroparesis.

This data will be used for research purposes only to determine the clinical impact of endoscopic treatments on gastroparesis. The physicians will also be able to better understand the patient's condition and disease process that may lead to improved standard of care and improved patient management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Referral for endoscopic treatment of Gastroparesis for symptom management

Exclusion Criteria:

* < 18 years of age
* Absence of gastroparesis based on scintigraphy studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As long as patients fall under the inclusion criteria and do not fall under exclusions, every patient can be considered. Patient must be declared safe to undergo procedure on individual basis from an evaluation from head doctor on study.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Change in Gastroparesis Cardinal Symptom Index (GCSI) from baseline to post G-POEM | 60 months span: baseline and assess change at 1 month, 3 month, 6 month, 12 month, 24 month, 36 month, 48 month & 60 months
  The Gastroparesis Cardinal Symptom Index (GCSI) is used for assessing severity of symptoms associated with gastroparesis. Patients are to score each of the 9 symptom criteria on 0 (None) to 5 (Very Severe) Likert Scale. The higher the score the more symptomatic from gastroparesis the patient is.
  Nausea or Vomiting (score 0-5 for each of the following 3 criteria)
  * Nausea
  * Retching
  * Vomiting Postprandial fullness or early satiety (score 0-5 for each of the following 4 criteria)
  * Stomach Fullness
  * Not able to finish a normal-sized meal
  * Feeling excessively full after meals
  * Loss of appetite Bloating (score 0-5 for each of the following 2 criteria)
  * Bloating
  * Stomach visibly larger
Assessment of Change in Patient Assessment of gastrointestinal disorders-symptom severity index (PAGI-SYM) score from baseline to post G-POEM | 60 months span: baseline and assess change at 1,3,6,12,24, 36,48 & 60 months
  Change in PAGI-Sym score: The PAGI-SYM is composed of 20 items and 6 subscales: heartburn/regurgitation (7 items), nausea/vomiting (3 items), postprandial fullness/early satiety (4 items), bloating (2 items), upper abdominal pain (2 items), and lower abdominal pain (2 items). Subscale scores are calculated by averaging across items comprising the subscale; scores vary from 0 (none or absent) to 5 (very severe)
Assessment of Change in G-POEM SF-36 Health Survey score from baseline to post G-POEM | baseline and assess change at 1,3,6,12,24,36,48 & 60 months
  Change in health belief questionnaire (SF-36) score: Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability and the higher scores indicate better health
Assessment of change in Gastric Emptying Scan (GES) (solid phase, 4 hour study) from baseline to post G-POEM | baseline; and assess change at 6, and 24 months
  we will track change in GES at 6 months and 24 months post G-POEM and compare to baseline. Normal GES should have under 5% at 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Al-Haddad, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Ichkhanian Y, Salame M, Wo JM, Nowak TV, Stainko S, Saito A, Siwiec RM, Kais A, Hwang JH, Li AA, Yang J, Broucek JR, Esfandyari T, Joseph S, Ujiki MB, Williams AE, Moremen J, Gouda Z, Schlachterman A, Hugova K, Martinek J, Geng CX, Podboy A, Wang AY, Lajin M, Gregor L, Miller PM, Al Bunni H, DeWitt JM, Al-Haddad M. A New International Scheme for the Classification and Management of Clinical Outcomes Post-gastric Peroral Endoscopic Myotomy. Clin Gastroenterol Hepatol. 2025 Dec;23(13):2477-2487.e1. doi: 10.1016/j.cgh.2025.03.022. Epub 2025 May 14. PMID 40378985
- [Derived] Salame M, Ichkhanian Y, Hadaki N, Wo JM, Stainko SA, Saito A, Siwiec RM, Nowak TV, Li A, Hwang JH, Yang J, Broucek J, Esfandyari T, Joseph S, Ujiki M, Williams AE, Moremen JR, Gouda Z, Schlachterman A, Hugova K, Martinek J, Geng CX, Podboy A, Wang AY, Lajin M, Miller P, Gregor L, Albunni H, Dewitt JM, Al-Haddad MA. Safety of same-day discharge after gastric peroral endoscopic myotomy in patients with refractory gastroparesis: an international multicenter study. Gastrointest Endosc. 2025 Oct;102(4):595-599.e1. doi: 10.1016/j.gie.2025.02.020. Epub 2025 Feb 19. PMID 39983999